CLINICAL TRIAL: NCT03155789
Title: Clinical Outcome After Lumbar Fusion for the Treatment of Chronic Low Back Pain
Brief Title: Clinical Outcome After Lumbar Fusion
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Gabriel C. Tender, MD, Clinical Professor, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: LSU-7270
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low Back Pain emanating from L4-5: 1. S TLIF at L4-5 (n=10)
  2. MI TLIF at L4-5 (n=10)
  3. XLIF at L4-5 (n=10)
  Interventions: Procedure: Lumbar Fusion
- Low Back Pain emanating from L5-S1: 1. S TLIF at L5-S1 (n=10)
  2. MI TLIF at L5-S1 (n=10)
  3. XLIF at L5-S1 (n=10)
  Interventions: Procedure: Lumbar Fusion
- Low Back Pain emanating from L4-5 and L5-S1: 1. S TLIF at L4-5 and L5-S1 (n=10)
  2. MI TLIF at L4-5 and L5-S1 (n=10)
  3. XLIF at L4-5 and L5-S1 (n=10)
  Interventions: Procedure: Lumbar Fusion

INTERVENTIONS:
Procedure: Lumbar Fusion — Standard Transforaminal Lumbar Interbody Fusion (S TLIF)
  Minimally Invasive Transforaminal Lumbar Interbody Fusion (MI TLIF)
  AxiaLIF Fusion

SUMMARY:
The main objective of this prospective study is to compare the clinical outcomes after lumbar fusion for chronic low back pain using the four techniques commonly employed in our surgical practice. Lumbar fusion stops motion at a painful vertebral segment, which can decrease back pain. The four techniques are standard transforaminal lumbar interbody fusion (S TLIF), minimally invasive transforaminal lumbar interbody fusion (MI TLIF), extreme lateral interbody fusion (XLIF), and axial lumbar interbody fusion (AxiaLIF). Each differ in where incisions are made and level of invasiveness; not all may be implemented in each surgical case. The four different techniques are all standard approaches with different advantages and have yet to be compared in efficacy for relieving chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Severe chronic low back pain (at least 7 out of 10 on the VAS scale).

  * Age: 25-65 years.
  * Pain duration at least 2 years.
  * The treating surgeon should interpret the pain as emanating from L4-S1.
  * The patient must have had unsuccessful maximal possible conservative (non surgical) treatment for at least one year.
  * Radiographic evidence (MRI, CT, CT-SPECT, and/or plain films) of degenerative changes ("spondylosis")

Exclusion Criteria:

* Psychiatric illness or evidence of emotional instability.

  * Previous spine surgery except for successful removal of a herniated disc more than 2 years before entering the study and with no persistent nerve root symptoms.
  * Specific radiologic findings, such as fractures, infection, inflammatory process, or neoplasm.
  * Obvious painful and disabling arthritic hip joints and anamnestic and radiologic signs of spinal stenosis.
  * Involvement in Workman's Comp or litigation.

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Each patient who is willing to participate in this study, signs informed consent, and complies with the inclusion/exclusion criteria will be enrolled in the study. Each patient will be enrolled chronologically on a patient enrollment log and given a patient number for the duration of the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Visual Analog Scale (VAS) | 2 weeks, 6 months, 1 year
  This is part of the Patient Questionnaire primary outcome measure. A Visual Analogue Scale (VAS) is a measurement instrument that measures the intensity or frequency of pain across a continuum of values.
Change from Baseline Prolo Functional and Economic Score | 2 weeks, 6 months, 1 year
  This is part of the Patient Questionnaire primary outcome measure. The Prolo Score is a 10-point scale consisting of only two questions evaluating the functional and economic status of the patient.
Change from Baseline Dallas Pain Questionnaire (DPQ) | 2 weeks, 6 months, 1 year
  This is part of the Patient Questionnaire primary outcome measure. The Dallas Pain Questionnaire (DPQ) assess the amount of chronic spine pain that affects the patient's daily and work-leisure activities, anxiety-depression, and social interest.
Change from Baseline Short Form 12 (SF-12) | 2 weeks, 6 months, 1 year
  This is part of the Patient Questionnaire primary outcome measure. The Short Form 12 (SF-12) was designed to measure the patient's functional health and well-being.
Change from Baseline Oswestry Disability Index (ODI) | 2 weeks, 6 months, 1 year
  This is part of the Patient Questionnaire primary outcome measure. The Oswestry Disability Index measures a patient's impairment and quality of life due to pain.

SECONDARY OUTCOMES:
Radiologic Fusion Rates | 6 months and 1 year
  Fusion rates will be evaluated by flexion-extension X-rays and CT imaging.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serban D, Calina N, Tender G. Standard versus Minimally Invasive Transforaminal Lumbar Interbody Fusion: A Prospective Randomized Study. Biomed Res Int. 2017;2017:7236970. doi: 10.1155/2017/7236970. Epub 2017 Jun 15. PMID 28698876